CLINICAL TRIAL: NCT02587182
Title: Effects of Dry Needling in Patients With Sleep Bruxism and Temporomandibular Disorders: a Prospective Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU-011
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Myofascial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dry needling (Experimental): Dry needling in the masseter and temporalis muscles
  Interventions: Device: Deep Dry needling

INTERVENTIONS:
Device: Deep Dry needling — The muscles were repeatedly perforated by rapidly inserting and partially withdrawing the needle from the myofascial trigger point, eliciting local twitch responses in some insertions

SUMMARY:
The objective of the present study was to assess the effectiveness of deep dry needling in the masseter and temporalis MTrPs on pain, pressure pain threshold (PPT), range of motion and disability in patients with sleep bruxism and myofascial temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myofascial temporomandibular disorders
* Diagnosis of myofascial trigger point
* Diagnosis of sleep bruxism

Exclusion Criteria:

* insurmountable fear of needles
* any systematic joint or muscle disease
* bleeding disorders or
* prior physical therapy treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain: visual analog scale, ranging from 0mm (no pain) to 100mm (worst imaginable pain). | 1 week
Pressure pain sensitivity: mechanical pressure algometer. | 1 week
Range of motion: distance between the upper and lower central dental incisors was measured with a millimeter ruler. | 1 week

REFERENCES:
- [Derived] Blasco-Bonora PM, Martin-Pintado-Zugasti A. Effects of myofascial trigger point dry needling in patients with sleep bruxism and temporomandibular disorders: a prospective case series. Acupunct Med. 2017 Mar;35(1):69-74. doi: 10.1136/acupmed-2016-011102. Epub 2016 Oct 3. PMID 27697769